CLINICAL TRIAL: NCT02383355
Title: Switch From an NNRTI or PI-based Regimen to a RAltegravir-based Regimen in Virologically Suppressed HIV-infected Patients: Effects on Platelet Reactivity, Platelet-monocyte Aggregation and the Inflammatory anD Thrombotic State of Monocytes
Brief Title: Effects of Raltegravir Based Regimen on Platelet Reactivity, Platelet-monocyte Aggregation and Immune Activation
Acronym: RAPID
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NL50681.091.14; 2014-1320 (Other: Local Ethical committee (Radboudumc))
Record Dates: First submitted 2015-01-23; First posted 2015-03-09 (Estimated); Results first posted 2019-01-10 (Actual); Last update posted 2019-01-10 (Actual); Status verified 2017-09

CONDITIONS: HIV
Keywords: Persistent immune activation; Platelet hyperreactivity
MeSH Terms: interventions — Raltegravir Potassium

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Switch group (Experimental): Raltegravir 400mg tablets administered twice daily together with continuation of their own backbone therapy for 10 weeks
  Interventions: Drug: Raltegravir
- Continuation group (Active Comparator): Individuals in the continuation group will continue the regimen, which consists of antiretroviral therapy as indicated in the inclusion criteria
  Interventions: Drug: Continuation of own regimen

INTERVENTIONS:
Drug: Raltegravir — Raltegravir 400mg tablets administered twice daily together with continuation of their own backbone therapy
  Other Names: Isentress
  Arms: Switch group
Drug: Continuation of own regimen — Continuation of own antiretroviral medication during the 10 weeks follow-up
  Arms: Continuation group

SUMMARY:
Cardiovascular disease (CVD) has emerged as a leading cause of morbidity and mortality in HIVinfected individuals. The precise mechanisms underlying this increased cardiovascular risk remain to be elucidated. Platelet hyperreactivity and increased platelet-monocyte aggregation (PMA) are found in HIVinfectedpatients and may contribute to the excess cardiovascular risk as platelets play a key role in the onset and progression of atherosclerosis and in acute cardiovascular events. In addition, HIV-infected individuals frequently suffer from persistent immune activation and inflammation. In a crosssectional study the investigators recently showed that individuals using a regimen containing the integrase inhibitor raltegravir have reduced platelet hyperreactivity and PMA compared to other antiretroviral regimens. Other recent studies showed that raltegravir is associated with decreased immune activation. Due to the inherent limitations of cross sectional studies, the investigators aim to expand our findings in an intervention study. The investigators will conduct a randomized control trial where the investigators switch patients to a integrase containing treatment regimen to assay possible changes in platelet function and persistent immune activation. Knowledge gathered in the proposed study can help understand and prevent cardiovascular disease in patients treated for a HIV infection by reducing platelet hyperreactivity and persistent immune activation.

DETAILED DESCRIPTION:
Rationale:

Cardiovascular disease (CVD) has emerged as a leading cause of morbidity and mortality in HIV-infected individuals. The precise mechanisms underlying this increased cardiovascular risk remain to be elucidated . Platelet hyperreactivity and increased platelet-monocyte aggregation (PMA) are found in HIV-infected patients and may contribute to the excess cardiovascular risk as platelets play a key role in the onset and progression of atherosclerosis and in acute cardiovascular events. In addition, HIV-infected individuals frequently suffer from persistent immune activation and inflammation. In a cross-sectional study the investigators recently showed that individuals using a regimen containing the integrase inhibitor raltegravir have reduced platelet hyperreactivity and PMA compared to other antiretroviral regimens. Other recent studies showed that raltegravir is associated with decreased immune activation. Due to the inherent limitations of cross sectional studies, the investigators aim to expand our findings in an intervention study.

Objective:

Investigate whether switch from a non-nucleoside reverse transcriptase inhibitor (NNRTI)- or protease inhibitor (PI)-based regimen to a raltegravir-based regimen results in reduced platelet reactivity, reduced platelet-leukocyte aggregate formation and pro-inflammatory status of monocytes.

Study design: Investigator initiated, single-center, open-label, randomized controlled trial in HIV-infected patients using a NNRTI- or PI-based regimen.

Study population:

Adult HIV-infected study participants with undetectable (<40 copies/mL) viral load receiving a standard backbone of two NRTI's (either tenofovir (TDF)/emtricitabine (FTC) or abacavir (ABC)/lamivudine (3TC)) with either a NNRTI (efavirenz (EFV) or rilpivirine (RPV)) or a boosted PI (Darunavir (DRV/r), atazanavir (ATZ/r) or Lopinavir (LPV/r)). After Sample size calculation two groups of 20 subjects will be enrolled.

Intervention:

Participants will be randomized (1:1) to continue the same ART regimen ("Continuation group") or to switch their NNRTI or PI to raltegravir ("Switch group") during 10 weeks.

Main study parameters/endpoints:

Primary parameter:

1. Platelet reactivity: platelet expression of the platelet activation marker CD62P (P-selectin) and activated fibrinogen receptor (αIIbβ3) upon stimulation with different platelet agonists.

Secondary parameters:

1. Platelet-leukocyte aggregates (eg. PMA).
2. Activation markers on T cells and monocytes.
3. Soluble (plasma) markers of platelet and monocyte activation.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Documented HIV-infection
* Age ≥ 18 years
* Willing to comply with the protocol requirements
* On stable antiretroviral therapy (ART) for ≥ 6 months at screening
* Undetectable plasma HIV viral load (<50 copies/mL) for at least 6 months
* CD4 cell count > 300 cells/mm3 at last measurement
* Current ART regimen at screening consisting of a backbone of two NRTI's (either TDF/FTC or ABC/3TC) with either a NNRTI (EFV or RPV) or a boosted PI (DRV/r, ATZ/r or LPV/r) and on this regimen for > 3 months
* If female and of childbearing potential using effective birth control methods

Exclusion Criteria:

* Use of platelet function inhibitors, such as aspirin and adenosine diphosphate (ADP) receptor antagonists
* Known hypersensitivity to raltegravir or any other component of the formulation
* Using any concomitant therapy disallowed as per summary of product characteristics (SPC) for the study drug
* Signs of symptoms of an active (opportunistic) infection other than HIV
* Active hepatitis B or C
* Estimated glomerular filtration rate (by MDRD) <50 ml/min
* Clinical or laboratory evidence of significantly decreased hepatic function, defined as alanine aminotransferase (ALAT) level > 2 upper limit of normal (ULN)
* History of suspected or proven virologic failure since ART initiation (HIV-1 RNA "blips" less than 500 copies per milliliter with subsequent suppression are allowed)
* Known genotypic resistance to any current ART component
* Prior use of single or dual NRTI-only regimens, or history of any ART not considered highly active by current standards.
* In females, pregnancy or breast feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-03-01 (Actual); Primary Completion 2016-03-31 (Actual); Study Completion 2017-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Quirijn de Mast, MD PhD, Principal Investigator — Radboud University (Radboudumc)

REFERENCES:
- [Result] Tunjungputri RN, Van Der Ven AJ, Schonsberg A, Mathan TS, Koopmans P, Roest M, Fijnheer R, Groot PG, de Mast Q. Reduced platelet hyperreactivity and platelet-monocyte aggregation in HIV-infected individuals receiving a raltegravir-based regimen. AIDS. 2014 Sep 10;28(14):2091-6. doi: 10.1097/QAD.0000000000000415. PMID 25265076
- [Derived] van der Heijden WA, van Crevel R, de Groot PG, Urbanus RT, Koenen HJPM, Bosch M, Keuter M, van der Ven AJ, de Mast Q. A switch to a raltegravir containing regimen does not lower platelet reactivity in HIV-infected individuals. AIDS. 2018 Nov 13;32(17):2469-2475. doi: 10.1097/QAD.0000000000001993. PMID 30134289

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Switch Group | Continuation Group
Started | 19 | 21
Completed | 17 | 21
Not Completed | 2 | 0
Not completed — Adverse Event | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Switch Group | Continuation Group | Total
Number analyzed (Participants) | 19 | 21 | 40
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 48 [43 to 54] | 49 [42 to 61] | 48 [43 to 58]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 18 | 21 | 39
Region of Enrollment [Number; unit: participants]
  Netherlands | 19 | 21 | 40

OUTCOME MEASURES:

1. Primary Outcome: Platelet Reactivity Measured by Expression of P-selectin (CD62p) and Fibrinogen Binding
Description: Platelet expression of the platelet activation marker CD62P (P-selectin) and of the activated fibrinogen receptor (αIIbβ3) through fibrinogen binding following stimulation with two concentrations of the platelet agonists ADP (adenosine diphosphate) and CRP-XL (crosslinked collagen related peptide). Difference between week 0 and week 10. Primary outcome is CD62p expression upon stimulation with ADP (power calculation based on this measure). Expression of both markers are expressed as MFI (Median fluorescence intensity) and measured by flowcytometry. Change after 10 weeks was calculated as a ratio between baseline and week 10.
Time Frame: Baseline and week 10
Population: Intention to treat, if week 10 is not available, week 4 was used for these individuals (n=2)
Measure: Median (Full Range); unit: Ratio
Arm/Group | Switch Group | Continuation Group
Number analyzed (Participants) | 19 | 21
Ratio
  ADP 125uM CD62p expression | 0.9 [0.49 to 1.14] | 0.96 [0.66 to 1.3]
  ADP 125uM Fibrinogen binding | 1 [0.37 to 2.8] | 0.99 [0.66 to 1.95]
  ADP 7.8uM CD62p expression | 0.88 [0.46 to 1.11] | 0.99 [0.690 to 1.32]
  ADP 7.8uM fibrinogen binding | 0.85 [0.39 to 2.13] | 1.02 [0.57 to 1.53]
  CRP (collagen) XL 655ng/ml CD62p expression | 0.95 [0.87 to 1.2] | 0.94 [0.68 to 1.28]
  CRP (collagen) XL 655ng/ml fibrinogen binding | 0.8 [0.48 to 1.77] | 0.8 [0.64 to 1.38]
  CRP (collagen) XL 27.33ng/ml CD62p expression | 0.87 [0.41 to 2.14] | 0.84 [0.33 to 1.84]
  CRP (collagen) XL 27.33 ng/ml fibrinogen binding | 0.88 [0.68 to 1.590] | 1.04 [0.41 to 1.59]

2. Secondary Outcome: Platelet-leukocyte Aggregates (Platelet Monocyte Complex Measured by Flow-cytometry)
Description: Platelet monocyte complex (PMCs) measured by flow-cytometry. % of CD61+ (platelet-marker) monocytes. Change after 10 weeks was calculated as a ratio between baseline and week 10.
Time Frame: Baseline and week 10
Measure: Median (Full Range); unit: ratio
Arm/Group | Switch Group | Continuation Group
Number analyzed (Participants) | 19 | 21
ratio | 0.95 [0.113 to 4.087] | 0.932 [0.198 to 3.604]

3. Secondary Outcome: T-cell Dysfunction (CD4-cells)
Description: Markers of persistent immune activation measured by flow cytometry (% of CD4-cells positive for CD38HLA-DR cells). Change after 10 weeks was calculated as a ratio between baseline and week 10.
Time Frame: Baseline and Week 10
Measure: Median (Full Range); unit: ratio
Arm/Group | Switch Group | Continuation Group
Number analyzed (Participants) | 19 | 21
ratio | 1.314 [0.309 to 10.78] | 1.016 [0.023 to 3.347]

4. Secondary Outcome: Circulating Levels of High Sensitive C-reactive Protein (Hs-CRP)
Description: Plasma levels of hs-CRP (ng/mL) measured by ELISA . Change in concentration was calculated as a ratio between baseline (week 0) and week 10.
Time Frame: Baseline and week 10
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Switch Group | Continuation Group
Number analyzed (Participants) | 19 | 18
ratio | 1.208 (0.895) | 1.103 (1.007)

5. Secondary Outcome: Persistent Immune Activation - Monocyte Subsets
Description: Monocyte subsets measured by flowcytometry. Classical monocytes (CD14+,CD16-), intermediate (CD14+CD16+), Non-classical (CD14dimCD16+). Reported values are change between baseline and week 10 and reported as ratio.
Time Frame: Baseline and week 10
Measure: Median (Full Range); unit: ratio
Arm/Group | Switch Group | Continuation Group
Number analyzed (Participants) | 19 | 21
ratio
  classical monocytes as % of total monocytes | 0.98 [0.777 to 1.095] | 0.998 [0.807 to 1.171]
  intermediate monocytes as % of total monocytes | 1.042 [0.325 to 2.923] | 0.979 [0.448 to 2.509]
  non-classical monocytes as % of total monocytes | 1 [0.567 to 2.128] | 1.089 [0.308 to 2.886]

ADVERSE EVENTS:
Arm/Group | Switch Group | Continuation Group
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/21
Other Adverse Events (participants affected / at risk) | 2/19 | 0/21
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Switch Group (N=19) | Continuation Group (N=21)
headache (Nervous system disorders) | 1 (1) | 0 (0) — headache
insomnia (Nervous system disorders) | 1 (1) | 0 (0) — insomnia

LIMITATIONS AND CAVEATS:
Even though our study was correctly powered for the primary outcome (platelet reactivity), the sample size gave us limited statistical power to explore all secondary objectives in detail and to include subanalyses exploring possible confounders.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes